CLINICAL TRIAL: NCT05511493
Title: Efficacy of Platelet-rich Plasma With Fractional Erbium-YAG Laser Versus With Microneedling in Localized Stable Vitiligo
Brief Title: Efficacy of PRP With Er-YAG Laser Versus With Microneedling in Localized Stable Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, aya marouf hameed aref, principal investigator, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRP in vitiligo
Record Dates: First submitted 2022-08-18; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Localized Vitiligo
MeSH Terms: interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: (Group A): Subjected to fractional erbium: yttrium-aluminum-garnet (Er: YAG) laser (FotonaXs Dynamis, Slovenia) with the energy of 1400 mJ in short pulse mode (SP) with spot size of 7 mm diameter, frequency of 3 Hz, and pixel 1. PRP is applied over the treated areas.
  (Group B): Subjected to microneedling using electronic dermapen device (Dr Pen Derma Pen Ultima A6®) which has a disposable head that personalized for each patient . The derma pen will penetrate the skin with variable depths ranging from 0.25 to 0.5 mm (not more than the depth of the epidermis). It will pass vertically over the vitiligo area in a circular pattern from the perilesional areas toward the depigmented center until pinpoint bleeding appears then the PRP is applied over the treated areas.
  * This procedure will be repeated every two weeks for six months.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fractional(Er: YAG) laser with platelet-rich plasma (Experimental): Subjected to fractional erbium: yttrium-aluminum-garnet (Er: YAG) laser (FotonaXs
  * Dynamis, Slovenia) with the energy of 1400 mJ in short pulse mode (SP) with spot size of 7 mm diameter, frequency of 3 Hz, and pixel 1. PRP is applied over the treated areas.This procedure will be repeated every two weeks for six months
  Interventions: Device: fractional Erbium-YAG laser
- Microneedling with platelet-rich plasma (Experimental): Subjected to microneedling using electronic dermapen device (Dr Pen Derma Pen Ultima A6®) which has a disposable head that personalized for each patient and sterilized after each session. The derma pen will penetrate the skin with variable depths ranging from 0.25 to 0.5 mm (not more than the depth of the epidermis). It will pass vertically over the vitiligo area in a circular pattern from the perilesional areas toward the depigmented center until pinpoint bleeding appears then the PRP is applied over the treated areas.
  - This procedure will be repeated every two weeks for six months.
  Interventions: Device: microneedling

INTERVENTIONS:
Device: fractional Erbium-YAG laser — Platelet-rich plasma with fractional Erbium-YAG laser in localized stable vitiligo
  Arms: fractional(Er: YAG) laser with platelet-rich plasma
Device: microneedling — Platelet-rich plasma with microneedling in localized stable vitiligo
  Arms: Microneedling with platelet-rich plasma

SUMMARY:
The aims of this study are to:- Compare the effect of fractional Erbium: YAG laser assisted delivery of platelet- rich plasma versus microneedling with platelet-rich plasma in the induction of skin repigmentation in localized stable vitiligo patients.

DETAILED DESCRIPTION:
Vitiligo is a depigmentation disease characterised by epidermal melanocyte death and melanin loss. It affects less than 0.1% to greater than 8% of the world's population. It is caused by a dynamic interplay between genetic and environmental risks that initiates an autoimmune attack on melanocytes in the skin. There are some treatment modalities, such as topical steroids, topical calcineurin inhibitors, excimer laser, narrowband-ultraviolet B therapy (NB-UVB), vitamin D,and non-cultured epidermal cell suspension (NCES).

One of the representative autogenous regenerative biomaterials is platelet-rich plasma (PRP) which contains moderate to high concentrations of platelets together with multiple biomolecules and moderate concentrations of leucocytes. Activated platelets can release autogenous growth factors that may initiate a signalling cascades and lead to numerous intracellular changes, promoting the proliferation, migration, and differentiation of stem cells and regulating local inflammation and immune responses.

Laser- assisted drug delivery (LADD) functions by creating focused zones of selective epidermal damage thereby rendering the dermis more accessible to topical medication.

Multiple lasers have been applied for the purpose of LADD, including ablative fractional carbon dioxide (CO2) and erbium-doped yttrium-aluminum-garnet (Er: YAG) lasers.

Microneedling (Mn) is a minimally invasive process in which many tiny needles penetrate the skin. It augments transdermal drug delivery (TDD) through the creation of pores in the stratum corneum. This technique is also believed to induce pigmentation by physically moving melanocytes with the needles into the vitiligo areas from the pigmented areas, so that they may serve as reservoirs for melanogenesis, also it induces microinflammation which stimulates the migration of keratinocytes and melanocytes that induces the release of cytokines and growth factors stimulating melanocytes at the periphery of vitiligo patches and their migration from pigmented to unpigmented areas.

ELIGIBILITY:
Inclusion Criteria:

- 1) Patients of both sexes with stable localized vitiligo: stable patches (should not have any increase or decrease in size or pigmentation for at least 3 months) .

2)Age between 10 - 60 years

Exclusion Criteria:

* 1)Acute or chronic infections. 2) Koebner phenomenon. 3) Contraindications to PRP injections:

  * Patients with blood or platelet abnormalities.
  * Patients taking anti-platelet drugs or anticoagulants.
  * Patients with a history of altered or abnormal fibroblast function, such as collagen diseases or myelofibrosis.

    4) We also excluded pregnant or lactating women. 5) All patients included had not received any local or systemic medication for at least 2 months before the study.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
percentage of skin repigmentation of localized stable vitiligo | six month
  according to Physician's Global Assessment [PGA] G4 (excellent: >75% repigmentation) G3 (very good: 50%-75% repigmentation) G2 (good: 25%-50% repigmentation)
  G1 (satisfactory: <25% repigmentation)
  G0 (poor: no repigmentation)
  The start of color and textural changes of skin will be examined every month. Assessment of pattern of repigmentation as marginal, perifollicular, diffuse and combined .

SECONDARY OUTCOMES:
Response to treatment | six month
  Response to treatment will be evaluated by photographing the patients and Physician's Global Assessment [PGA] at the baseline before the treatment and monthly after starting the treatment to detect the correlation between the degrees of repigmentation in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Hassan M Ibrahim, Ass. Prof, Study Director — southvalley university; Eisa M Hegazy, Ass. Prof, Study Director — southvalley university; Soheir ab Ali, Dr., Study Director — southvalley university

REFERENCES:
- [Background] Jin Y, Andersen G, Yorgov D, Ferrara TM, Ben S, Brownson KM, Holland PJ, Birlea SA, Siebert J, Hartmann A, Lienert A, van Geel N, Lambert J, Luiten RM, Wolkerstorfer A, Wietze van der Veen JP, Bennett DC, Taieb A, Ezzedine K, Kemp EH, Gawkrodger DJ, Weetman AP, Koks S, Prans E, Kingo K, Karelson M, Wallace MR, McCormack WT, Overbeck A, Moretti S, Colucci R, Picardo M, Silverberg NB, Olsson M, Valle Y, Korobko I, Bohm M, Lim HW, Hamzavi I, Zhou L, Mi QS, Fain PR, Santorico SA, Spritz RA. Genome-wide association studies of autoimmune vitiligo identify 23 new risk loci and highlight key pathways and regulatory variants. Nat Genet. 2016 Nov;48(11):1418-1424. doi: 10.1038/ng.3680. Epub 2016 Oct 10. PMID 27723757
- [Background] Alikhan A, Felsten LM, Daly M, Petronic-Rosic V. Vitiligo: a comprehensive overview Part I. Introduction, epidemiology, quality of life, diagnosis, differential diagnosis, associations, histopathology, etiology, and work-up. J Am Acad Dermatol. 2011 Sep;65(3):473-491. doi: 10.1016/j.jaad.2010.11.061. PMID 21839315
- [Background] Rashighi M, Harris JE. Vitiligo Pathogenesis and Emerging Treatments. Dermatol Clin. 2017 Apr;35(2):257-265. doi: 10.1016/j.det.2016.11.014. PMID 28317534
- [Background] Whitton M, Pinart M, Batchelor JM, Leonardi-Bee J, Gonzalez U, Jiyad Z, Eleftheriadou V, Ezzedine K. Evidence-based management of vitiligo: summary of a Cochrane systematic review. Br J Dermatol. 2016 May;174(5):962-9. doi: 10.1111/bjd.14356. Epub 2016 Mar 25. PMID 26686510
- [Background] Chen J, Wan Y, Lin Y, Jiang H. The application of platelet-rich plasma for skin graft enrichment: A meta-analysis. Int Wound J. 2020 Dec;17(6):1650-1658. doi: 10.1111/iwj.13445. Epub 2020 Jul 7. PMID 32633467
- [Background] Lee WR, Shen SC, Al-Suwayeh SA, Li YC, Fang JY. Erbium:YAG laser resurfacing increases skin permeability and the risk of excessive absorption of antibiotics and sunscreens: the influence of skin recovery on drug absorption. Toxicol Lett. 2012 Jun 1;211(2):150-8. doi: 10.1016/j.toxlet.2012.03.797. Epub 2012 Mar 29. PMID 22483991
- [Background] Zaleski-Larsen LA, Fabi SG. Laser-Assisted Drug Delivery. Dermatol Surg. 2016 Aug;42(8):919-31. doi: 10.1097/DSS.0000000000000556. PMID 27191783
- [Background] Hou A, Cohen B, Haimovic A, Elbuluk N. Microneedling: A Comprehensive Review. Dermatol Surg. 2017 Mar;43(3):321-339. doi: 10.1097/DSS.0000000000000924. PMID 27755171
- [Background] Vandervoort J, Ludwig A. Microneedles for transdermal drug delivery: a minireview. Front Biosci. 2008 Jan 1;13:1711-5. doi: 10.2741/2794. PMID 17981662
- [Background] Wassef C, Lombardi A, Khokher S, Rao BK. Vitiligo surgical, laser, and alternative therapies: a review and case series. J Drugs Dermatol. 2013 Jun 1;12(6):685-91. PMID 23839187
- [Derived] Abdel-Hamid S, Ibrahim HM, Hameed AM, Hegazy EM. Effectiveness of fractional erbium-YAG laser, microneedling, platelet-rich plasma in localized stable vitiligo patients: randomized clinical trial. Arch Dermatol Res. 2024 Jun 15;316(7):399. doi: 10.1007/s00403-024-03035-8. PMID 38878236